CLINICAL TRIAL: NCT03264859
Title: Neutrophil Gelatinase-associated Lipocalin (NGAL) and Its Association With the No-reflow Phenomenon in ST-elevation Myocardial Infarction
Brief Title: NGAL and Its Association With the No-reflow Phenomenon in ST-elevation Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Zotal Inc. (Unknown)
Responsible Party: Principal Investigator, Dr. Shlomi Matetzky, Head, Intensive Care Care Unit, Sheba Medical Center
Other Study IDs: SHEBA-17-4157-SM-CTIL
Record Dates: First submitted 2017-08-14; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: No-Reflow Phenomenon; STEMI - ST Elevation Myocardial Infarction
Keywords: NGAL; STEMI; no-reflow; PCI (Percutaneous Coronary Intervention)
MeSH Terms: conditions — No-Reflow Phenomenon; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: NGAL levels early and post STEMI — NGAL levels early and post ST elevation MI (STEMI)

SUMMARY:
The aim of this study is to investigate the association between NGAL plasma levels in ST-elevation myocardial infarction and the no-reflow phenomenon, adverse events during hospitalization and at 30-day follow-up.

DETAILED DESCRIPTION:
Neutrophil Gelatinase-associated Lipocalin (NGAL) is a acute phase protein which is elevated in conditions like acute kidney injury and myocardial infarction. When a coronary artery is occluded, detrimental changes occur in myocardial vessels. After relief of the occlusion, blood flow to the heart may still be impeded, a phenomenon known as "no-reflow". Data is lacking on factors associated with early detection of patients at risk for this phenomenon, and early stratification of this group seems vital since the no-reflow phenomenon is associated with worse outcomes. The investigators hypothesized that there might be an association between higher NGAL levels and the occurrence of no-flow findings, and that NGAL might serve as a marker of worse prognosis in this population. The investigators also hypothesized that NGAL levels might serve as a marker of early acute kidney injury and that there might be specific patterns of NGAL levels over time in different subsets of patients. The aim of the study is to determine the association between NGAL levels at admission and during the first days after a ST-elevation myocardial infarction, the occurrence of the no-reflow phenomenon, the extent of myocardial damage ascertained by cardiac imaging techniques (echocardiography and cardiac resonance imaging). Data regarding patients' clinical, laboratory, electrocardiogram, coronary angiography and percutaneous coronary intervention, in-hospital and 30-day follow-up after discharge will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old presenting with ST-elevation myocardial infarction and undergoing urgent coronary angiography with or without PCI.
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Inability to sign written informed consent.
* Chronic renal failure (eGFR < 30 ml/min/1.73m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Sheba Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
No-reflow phenomenon after STEMI | During hospitalization
  No-reflow phenomenon as defined by electrocardiographic, angiographic and cardiac magnetic resonance imaging criteria.

SECONDARY OUTCOMES:
In-hospital MACE(major adverse cardiac events) | Average day 5 of hospitalization and before discharge
  In-hospital MACE
30-day MACE | 30-day follow-up
  30-day MACE
Serial creatinine level | On admission and at fixed time intervals (first 3 hours after admission, 12 hours, 24 hours and every 24 hours or before if indicated)
  Creatinine levels as a maker of acute kidney injury reported in mg/dl
The need for renal replacement therapy after STEMI | In-hospital (usually 5 days)
  Patients started on hemodyalisis due to acute kidney injury during the index hospitalization
Recurrent hospitalization | 30 days
  Recurrent hospitalization at 30 days after the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Shlomi Matetzky, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Cardiac Intensive Care Unit, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kjeldsen L, Johnsen AH, Sengelov H, Borregaard N. Isolation and primary structure of NGAL, a novel protein associated with human neutrophil gelatinase. J Biol Chem. 1993 May 15;268(14):10425-32. PMID 7683678
- [Background] Xu SY, Carlson M, Engstrom A, Garcia R, Peterson CG, Venge P. Purification and characterization of a human neutrophil lipocalin (HNL) from the secondary granules of human neutrophils. Scand J Clin Lab Invest. 1994 Aug;54(5):365-76. doi: 10.3109/00365519409088436. PMID 7997842
- [Background] Mishra J, Dent C, Tarabishi R, Mitsnefes MM, Ma Q, Kelly C, Ruff SM, Zahedi K, Shao M, Bean J, Mori K, Barasch J, Devarajan P. Neutrophil gelatinase-associated lipocalin (NGAL) as a biomarker for acute renal injury after cardiac surgery. Lancet. 2005 Apr 2-8;365(9466):1231-8. doi: 10.1016/S0140-6736(05)74811-X. PMID 15811456
- [Background] Leclercq A, Houard X, Philippe M, Ollivier V, Sebbag U, Meilhac O, Michel JB. Involvement of intraplaque hemorrhage in atherothrombosis evolution via neutrophil protease enrichment. J Leukoc Biol. 2007 Dec;82(6):1420-9. doi: 10.1189/jlb.1106671. Epub 2007 Sep 7. PMID 17827339
- [Background] Zografos T, Haliassos A, Korovesis S, Giazitzoglou E, Voridis E, Katritsis D. Association of neutrophil gelatinase-associated lipocalin with the severity of coronary artery disease. Am J Cardiol. 2009 Oct 1;104(7):917-20. doi: 10.1016/j.amjcard.2009.05.023. PMID 19766756
- [Background] Wagener G, Jan M, Kim M, Mori K, Barasch JM, Sladen RN, Lee HT. Association between increases in urinary neutrophil gelatinase-associated lipocalin and acute renal dysfunction after adult cardiac surgery. Anesthesiology. 2006 Sep;105(3):485-91. doi: 10.1097/00000542-200609000-00011. PMID 16931980
- [Background] Bachorzewska-Gajewska H, Malyszko J, Sitniewska E, Malyszko JS, Dobrzycki S. Neutrophil-gelatinase-associated lipocalin and renal function after percutaneous coronary interventions. Am J Nephrol. 2006;26(3):287-92. doi: 10.1159/000093961. Epub 2006 Jun 13. PMID 16772710
- [Background] Lindberg S, Jensen JS, Hoffmann S, Iversen AZ, Pedersen SH, Biering-Sorensen T, Galatius S, Flyvbjerg A, Mogelvang R, Magnusson NE. Plasma Neutrophil Gelatinase-Associated Lipocalin Reflects Both Inflammation and Kidney Function in Patients with Myocardial Infarction. Cardiorenal Med. 2016 May;6(3):180-90. doi: 10.1159/000443846. Epub 2016 Feb 25. PMID 27275154
- [Background] Morishima I, Sone T, Okumura K, Tsuboi H, Kondo J, Mukawa H, Matsui H, Toki Y, Ito T, Hayakawa T. Angiographic no-reflow phenomenon as a predictor of adverse long-term outcome in patients treated with percutaneous transluminal coronary angioplasty for first acute myocardial infarction. J Am Coll Cardiol. 2000 Oct;36(4):1202-9. doi: 10.1016/s0735-1097(00)00865-2. PMID 11028471
- [Background] Aksan G, Soylu K, Aksoy O, Ozdemir M, Yanik A, Yuksel S, Gedikli O, Gulel O, Sahin M. The relationship between neutrophil gelatinase-associated lipocalin levels and the slow coronary flow phenomenon. Coron Artery Dis. 2014 Sep;25(6):505-9. doi: 10.1097/MCA.0000000000000121. PMID 24801557
- [Background] Helanova K, Littnerova S, Kubena P, Ganovska E, Pavlusova M, Kubkova L, Jarkovsky J, Pavkova Goldbergova M, Lipkova J, Gottwaldova J, Kala P, Toman O, Dastych M, Spinar J, Parenica J. Prognostic impact of neutrophil gelatinase-associated lipocalin and B-type natriuretic in patients with ST-elevation myocardial infarction treated by primary PCI: a prospective observational cohort study. BMJ Open. 2015 Oct 5;5(10):e006872. doi: 10.1136/bmjopen-2014-006872. PMID 26438132
- [Background] Akcay AB, Ozlu MF, Sen N, Cay S, Ozturk OH, Yalcn F, Bilen P, Kanat S, Karakas MF, Isleyen A, Demir AD, Sogut S, Covic A, Kanbay M. Prognostic significance of neutrophil gelatinase-associated lipocalin in ST-segment elevation myocardial infarction. J Investig Med. 2012 Feb;60(2):508-13. doi: 10.2310/JIM.0b013e31823e9d86. PMID 22222228
- [Background] Durante A, Laricchia A, Benedetti G, Esposito A, Margonato A, Rimoldi O, De Cobelli F, Colombo A, Camici PG. Identification of High-Risk Patients After ST-Segment-Elevation Myocardial Infarction: Comparison Between Angiographic and Magnetic Resonance Parameters. Circ Cardiovasc Imaging. 2017 Jun;10(6):e005841. doi: 10.1161/CIRCIMAGING.116.005841. PMID 28592591